CLINICAL TRIAL: NCT01568463
Title: What is the Maximal Effective Distance for Interscalene Block?
Brief Title: Distance for Interscalene Block
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0806-A
Record Dates: First submitted 2012-03-06; First posted 2012-04-02 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Regional Anesthesia; Inter Scalene Block; Post Operative Analgesia
Keywords: Inter-scalene Block; Regional Anesthesia; shoulder surgeries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Patients experience significant postoperative pain following shoulder surgery, Single shot interscalene block is used in ambulatory shoulder surgery for its advantages that include significant reduction in acute pain and analgesic requirements, prolonged time to first analgesic request, decreased incidence of nausea, as well as earlier hospital discharge.The process of nerve block requires several needle passes, with each of them being at risk of causing nerve injury either by direct trauma or intraneural injection even with the use of the ultrasound. These facts raised concerns and several authors stated that maybe the anesthesiologists should be more careful, keep a safe distance from the nerve, and inject the local anesthetics into fascial planes containing the nerve and not attempt to place the needle in close proximity to the nerve. This study is designed to determine the maximal effective distance away from the nerve for the injection to be effective.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-85 years of age, inclusive
* surgery less than 3 hours

Exclusion Criteria:

* contraindications to brachial plexus block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
* existing neurological deficit in the area to be blocked
* pregnancy
* history of neck surgery or radiotherapy
* severe respiratory disease
* inability to understand the informed consent and demands of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing shoulder surgery (shoulder arthroscopy or open shoulder surgery)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-01-24 (Actual); Study Completion 2014-03-26 (Actual)

PRIMARY OUTCOMES:
Success of the inter-scalene block at 20 minutes after injection at a specific distance of the needle tip from the outer sheeth of the nerve | 20 mins

SECONDARY OUTCOMES:
The onset time of sensory and motor block | the block success will be assessed for each patient every 5 min for 20 mins in the block room beginning when the needle exits the skin
The proportion of inadequate and failed blocks. | the block success will be assessed for each patient every 5 min for 20 mins in the block room beginning when the needle exits the skin
The duration of block, defined as the time from the completion of block performance to the time of the request for the first postoperative analgesic. | during the first 24 hours post operative
The amount of pain and level of satisfaction, | every 30 minutes starting at post anesthesia care unit admission till 120 minutes
The presence of a Claude-Bernard-Horner Syndrome | up to 24 hours post operative
The presence of hoarseness. | up to 24 hours post operative
The presence of other complications such as hematoma, infection, pneumothorax. | up to 24 hours post operative and 7 days post op

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada